CLINICAL TRIAL: NCT03395275
Title: Intrathecal Morphine Microdose Method Sensory Changes: A Pilot Study
Brief Title: Intrathecal Morphine Microdose Method Sensory Changes
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of recruitment and funding
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 17-0245
Record Dates: First submitted 2017-12-05; First posted 2018-01-10 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Analgesic Drug Dependence; Sensory Disorders; Chronic Pain
MeSH Terms: conditions — Sensation Disorders; Chronic Pain | interventions — Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: The study will be a non-randomized prospective trial. Participants will be selected for microdose intrathecal pump therapy by their pain physicians. Eligible participants will undergo an opioid taper by their physicians, and sensory tests will be carried out in the various stages of the intrathecal microdose treatment process (pre-taper, mid-taper, post-taper and post-implant phase).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intrathecal Pump Therapy Participants (Experimental): Patients eligible for intrathecal pump therapy will undergo quantitative sensory tests and surveys during various stages of the treatment process.
  Interventions: Behavioral: Quantitative Sensory Tests; Behavioral: surveys

INTERVENTIONS:
Behavioral: Quantitative Sensory Tests — Three testing modalities will be utilized for this study:
  1. Hot threshold test: The hot threshold method we will be utilizing has been described in the literature with good reproducibility and reliability. We will be using a similar system and have reproduced the program using a non-invasive device.
  2. Cold threshold test: the same non-invasive device will be used to test cold detection and pain threshold levels. This method is previously described.
  3. Pressure threshold: Mechanical testing (pressure pain threshold) will be assessed utilizing an algometer. We have used this method in a previous study and published results.
Behavioral: surveys — surveys including anxiety, depression, pain behavior, fatigue, pain interference, physical function, sleep disturbance, self-efficacy, satisfaction roles

SUMMARY:
Following the retrospective study on the effectiveness of the microdose method of intrathecal morphine therapy, the investigators are interested in measuring the sensory changes at 4 time points during the microdose method. The microdose method involves weaning the patient off oral opioids and maintaining an opioid-free period prior to initiating a very low opioid dose in intrathecal therapy. The microdose method is a standard of care. The study involves measuring sensory changes to hot, cold, and pressure. Data collection will be performed at regularly scheduled clinic visits, examining range of doses, pain scores,dose escalations, quantifiable psychosocial factors ( not captured in previous retrospective study), and changes in sensory thresholds.

DETAILED DESCRIPTION:
The use of intrathecal drug delivery systems for the management of chronic non-cancer pain has been in practice for over 30 years. A recently published study from the University of Texas Medical Branch performed a retrospective review on the morphine microdose method in community-based clinics. The goal of the study was to examine the morphine microdose method in an outpatient setting and assess success of therapy, pain scores and dose escalation. Patients were successfully weaned off their systemic opioids, maintained in an opioid-free period for 4-6 weeks, and then underwent a microdose trial and implantation. The majority of patients were successfully managed on morphine monotherapy, with a significant reduction in pain scores, and dose escalations comparable to prior studies. No prospective studies have examined the microdose method in correlation with changes in pain sensitivity.

Several studies have looked at the use of various pain testing models to investigate the effects of chronic opioid therapy and changes in pain perception. A systematic review of the literature identified clinical studies incorporating measures of hyperalgesia in patients on chronic opioid therapy. This review was aimed at finding the optimal testing modality to evaluate pain threshold and tolerance to external stimuli, including mechanical (pressure, touch, injection), thermal (cold/heat), and electrical. Although the results did not reveal any one method with sufficient power, several prospective studies evaluating hyperalgesia with heat pain ratings have shown some promising results; two studies revealing significant changes in heat responses for opioid treatment groups, and one study demonstrating lower heat pain perception values following an opioid taper. The latter study of research pertaining to pain sensitivity changes following an opioid taper is lacking, and only recently was a study performed investigating changes in pressure threshold following transition from full mu agonist to buprenorphine. Little is known at this juncture how pain thresholds change due to opioid dose changes and/or route of delivery changes such as oral to intrathecal routes.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75
* Selected for microdose Intrathecal pump therapy by their pain physician
* Chronic pain for at least 3 months
* Willing to cooperate with all study procedures

Exclusion Criteria:

* Presence of cancer
* Age less than 18 years old or greater than 75
* Current intrathecal therapy and/or with multiple intrathecal drugs (such as other opioids, local anesthetics, muscle relaxants)
* Medical conditions (myocardial infarction within the last year, uncontrolled diabetes, autoimmune disease
* Recent history of alcohol or substance abuse in the last 5 years

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-10-08 (Actual); Primary Completion 2023-02-03 (Actual); Study Completion 2023-02-03 (Actual)

PRIMARY OUTCOMES:
Heat threshold measurements | 2 years
  Heat threshold measurements (degrees Celsius) will be obtained using a pen-shaped temperature probe. Tests will be performed on a designated painful and non-painful body surface. Testing will completed when patient reports numeric pain rating of 5 or greater, or at a temperature >49 degrees Celsius.
Cold threshold measurements | 2 years
  Cold threshold measurements (degrees Celsius) will be obtained using a pen-shaped temperature probe. Tests will be performed on a designated painful and non-painful body surface. Testing will be completed when patient reports discomfort with cold stimulus, or if probe temperature reaches 0 degrees Celsius.
Pressure threshold measurements | 2 years
  Pressure threshold measurements (Newtons) will be obtained using a hand-held algometer. Tests will be performed on a designated painful and non-painful body surface. Testing will be completed when patient reports discomfort with pressure stimulus, or if pressure exceeds 60 Newtons.

SECONDARY OUTCOMES:
Demographic Evaluation - Pain History | 2 years
  To describe the patient population and to evaluate patient factors, which predict successful trials. The investigators will do a chart review of one year prior to start of the trial to examine the pain history.
Demographic Evaluation - Medical History | 2 years
  To describe the patient population and to evaluate patient factors, which predict successful trials. The investigators will do a chart review of one year prior to start of the trial to examine the medical history.
Demographic Evaluation - Body Mass Index | 2 years
  To describe the patient population and to evaluate patient factors, which predict successful trials. The investigators will collect data on body mass index.
Demographic Evaluation - Gender | 2 years
  To describe the patient population and to evaluate patient factors, which predict successful trials. The investigators will collect data on gender.
Demographic Evaluation - Surgical History | 2 years
  To describe the patient population and to evaluate patient factors, which predict successful trials. We will do a chart review of one year prior to start of the trial to examine the surgical history.
Demographic Evaluation - Age | 2 years
  To describe the patient population and to evaluate patient factors, which predict successful trials. The investigators will collect data on patient age.
Demographic Evaluation - Social History | 2 years
  To describe the patient population and to evaluate patient factors, which predict successful trials. We will do a chart review of one year prior to start of the trial to examine the social history.
Demographic Evaluation - Urine Drug Tests | 2 years
  To describe the patient population and to evaluate patient factors, which predict successful trials. We will do a chart review of one year prior to start of the trial to examine the urine drug tests
Demographic Evaluation - Numeric Pain Scale Scores | 2 years
  To describe the patient population and to evaluate patient factors, which predict successful trials. We will do a chart review of one year prior to start of the trial to examine numeric pain scale scores.
surveys - Anxiety | 2 years
  Patient-Reported Outcomes Measurement Information System survey on anxiety will be administered at the subject's initial, halfway and end of their evaluations. The results from the surveys will be aggregated and compared to other participants' responses.
surveys - Depression | 2 years
  Patient-Reported Outcomes Measurement Information System survey on depression will be administered at the subject's initial, halfway and end of their evaluations. The results from the surveys will be aggregated and compared to other participants' responses.
surveys - Pain Behavior | 2 years
  Patient-Reported Outcomes Measurement Information System survey on pain behavior will be administered at the subject's initial, halfway and end of their evaluations. The results from the surveys will be aggregated and compared to other participants' responses.
surveys - Fatigue | 2 years
  Patient-Reported Outcomes Measurement Information System survey on fatigue will be administered at the subject's initial, halfway and end of their evaluations. The results from the surveys will be aggregated and compared to other participants' responses.
surveys - Pain Interference | 2 years
  Patient-Reported Outcomes Measurement Information System survey on pain interference will be administered at the subject's initial, halfway and end of their evaluations. The results from the surveys will be aggregated and compared to other participants' responses.
surveys - Physical Function | 2 years
  Patient-Reported Outcomes Measurement Information System survey on physical function will be administered at the subject's initial, halfway and end of their evaluations. The results from the surveys will be aggregated and compared to other participants' responses.
surveys - Sleep Disturbance | 2 years
  Patient-Reported Outcomes Measurement Information System survey on sleep disturbance will be administered at the subject's initial, halfway and end of their evaluations. The results from the surveys will be aggregated and compared to other participants' responses.

CONTACTS AND LOCATIONS:
Overall Officials: Denise M Wilkes, MD, Principal Investigator — Associate Professor

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wallace M, Yaksh TL. Long-term spinal analgesic delivery: a review of the preclinical and clinical literature. Reg Anesth Pain Med. 2000 Mar-Apr;25(2):117-57. doi: 10.1053/rapm.2000.0250117. No abstract available. PMID 10746527
- [Background] Wilkes DM, Orillosa SJ, Hustak EC, Williams CG, Doulatram GR, Solanki DR, Garcia EA, Huang LM. Efficacy, Safety, and Feasibility of the Morphine Microdose Method in Community-Based Clinics. Pain Med. 2018 Sep 1;19(9):1782-1789. doi: 10.1093/pm/pnx132. PMID 29016893
- [Background] Hamza M, Doleys D, Wells M, Weisbein J, Hoff J, Martin M, Soteropoulos C, Barreto J, Deschner S, Ketchum J. Prospective study of 3-year follow-up of low-dose intrathecal opioids in the management of chronic nonmalignant pain. Pain Med. 2012 Oct;13(10):1304-13. doi: 10.1111/j.1526-4637.2012.01451.x. Epub 2012 Jul 30. PMID 22845187
- [Background] Grider JS, Harned ME, Etscheidt MA. Patient selection and outcomes using a low-dose intrathecal opioid trialing method for chronic nonmalignant pain. Pain Physician. 2011 Jul-Aug;14(4):343-51. PMID 21785477
- [Background] Pud D, Cohen D, Lawental E, Eisenberg E. Opioids and abnormal pain perception: New evidence from a study of chronic opioid addicts and healthy subjects. Drug Alcohol Depend. 2006 May 20;82(3):218-23. doi: 10.1016/j.drugalcdep.2005.09.007. Epub 2005 Oct 17. PMID 16229972
- [Background] Chu LF, D'Arcy N, Brady C, Zamora AK, Young CA, Kim JE, Clemenson AM, Angst MS, Clark DJ. Analgesic tolerance without demonstrable opioid-induced hyperalgesia: a double-blinded, randomized, placebo-controlled trial of sustained-release morphine for treatment of chronic nonradicular low-back pain. Pain. 2012 Aug;153(8):1583-1592. doi: 10.1016/j.pain.2012.02.028. Epub 2012 Jun 16. PMID 22704854
- [Background] Krishnan S, Salter A, Sullivan T, Gentgall M, White J, Rolan P. Comparison of pain models to detect opioid-induced hyperalgesia. J Pain Res. 2012;5:99-106. doi: 10.2147/JPR.S27738. Epub 2012 Apr 27. PMID 22570562
- [Background] Wasserman RA, Hassett AL, Harte SE, Goesling J, Malinoff HL, Berland DW, Zollars J, Moser SE, Brummett CM. Pressure Pain Sensitivity in Patients With Suspected Opioid-Induced Hyperalgesia. Reg Anesth Pain Med. 2015 Nov-Dec;40(6):687-93. doi: 10.1097/AAP.0000000000000315. PMID 26469365
- [Background] Katz NP, Paillard FC, Edwards RR. Review of the performance of quantitative sensory testing methods to detect hyperalgesia in chronic pain patients on long-term opioids. Anesthesiology. 2015 Mar;122(3):677-85. doi: 10.1097/ALN.0000000000000530. PMID 25437498
- [Background] Suzan E, Eisenberg E, Treister R, Haddad M, Pud D. A negative correlation between hyperalgesia and analgesia in patients with chronic radicular pain: is hydromorphone therapy a double-edged sword? Pain Physician. 2013 Jan;16(1):65-76. PMID 23340535
- [Background] Hooten WM, Mantilla CB, Sandroni P, Townsend CO. Associations between heat pain perception and opioid dose among patients with chronic pain undergoing opioid tapering. Pain Med. 2010 Nov;11(11):1587-98. doi: 10.1111/j.1526-4637.2010.00962.x. Epub 2010 Oct 1. PMID 21029354
- [Background] Wasserman RA, Hassett AL, Harte SE, Goesling J, Malinoff HL, Berland DW, Zollars J, Moser SE, Brummett CM. Pressure sensitivity and phenotypic changes in patients with suspected opioid-induced hyperalgesia being withdrawn from full mu agonists. J Nat Sci. 2017 Feb;3(2):e319. PMID 28361126
- [Background] Dyck PJ, Zimmerman IR, Johnson DM, Gillen D, Hokanson JL, Karnes JL, Gruener G, O'Brien PC. A standard test of heat-pain responses using CASE IV. J Neurol Sci. 1996 Mar;136(1-2):54-63. doi: 10.1016/0022-510x(95)00277-9. PMID 8815179
- [Background] Wright A, Benson HAE, Will R, Moss P. Cold Pain Threshold Identifies a Subgroup of Individuals With Knee Osteoarthritis That Present With Multimodality Hyperalgesia and Elevated Pain Levels. Clin J Pain. 2017 Sep;33(9):793-803. doi: 10.1097/AJP.0000000000000458. PMID 27898461
- [Background] Wilkes D, Martinello C, Medeiros FA, Babazade R, Hurwitz E, Khanjee N, Iyer PS, Leary P, Vadhera RB. Ultrasound-determined landmarks decrease pressure pain at epidural insertion site in immediate post-partum period. Minerva Anestesiol. 2017 Oct;83(10):1034-1041. doi: 10.23736/S0375-9393.17.11782-7. Epub 2017 Apr 11. PMID 28402092